CLINICAL TRIAL: NCT07165119
Title: The Effect of the Clinical Pilates, Nurse Coaching and Peer Group Work Approach on General Health Parameters in the Elderly With Diabetes: A Randomized Controlled
Brief Title: The Effect of the Interdisciplinary Care Approach on General Health Parameters in Older Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Kutay Kaslı, Dr, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 435; Kutay Kaşlı (Other: Çankırı Karatekin University)
Record Dates: First submitted 2025-08-27; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: elderly diabetic; nurse coaching; Pilates; interdisciplinary care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study was carried out as a single-blind, 4-arm randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors conducted initial and post-treatment assessments of participants in the study. Training was carried out on different days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Interdisciplinary group (Experimental): For 12 weeks, 3 times interdisciplinary treatment for 12 participants.
  Interventions: Other: Interdisciplinary group
- Nurse Coaching group (Active Comparator): nurse coaching for 12 weeks lasting 45 minutes once a week for 12 participants.
  Interventions: Other: Nurse Coaching group
- Clinical Pilates group (Active Comparator): Clinical Pilates For 12 weeks, 3 times exercise for 12 participants.
  Interventions: Other: Clinical Pilates Group
- Control group (No Intervention): Control group: 12 week waiting list for 12 participants.

INTERVENTIONS:
Other: Interdisciplinary group — For 12 weeks, the subjects in the interdisciplinary group participated in 45 minutes of clinical Pilates three times a week, as in the clinical Pilates group, and 45 minutes of nurse coaching once a week, as in the nurse coaching group.
  Arms: Interdisciplinary group
Other: Clinical Pilates Group — Clinical Pilates was applied by a certified physiotherapist for 12 consecutive weeks. with 45-minute sessions 3 times a week and was delivered to small groups of participants (3-5). The Pilates program has been developed in accordance with the extant literature to cultivate strength, balance, and coordination in a range of body positions, including the supine, seated, kneeling, and standing positions. Participants were instructed to perform each movement with control and precision, focusing on proper breathing patterns (exhaling during flexion, inhaling during extension) and engaging their core muscles throughout the exercise The load level and progression were determined using the Borg CR10 scale: Borg ≤ 2 = light load; Borg > 2 - < 5 = moderate load; Borg ≥ 5 - < 7 = heavy load; Borg ≥ 7 = near-maximum load. During the sessions, the effort level was generally maintained at a moderate intensity (Borg 3-4). Each time the intensity of the exercise was changed, the new loa
  Arms: Clinical Pilates group
Other: Nurse Coaching group — Training and follow-up was carried out with nurse coaching for 12 weeks lasting 45 minutes once a week .
  Arms: Nurse Coaching group

SUMMARY:
The aim of the study was evaluation of the effect of the clinical Pilates, nurse coaching and Peer group work Approach on General Health Parameters in older adults with Diabetes. This study was conducted as a single-blind, 4-arm, single-randomized and controlled study to estimate the effect of clinical Pilates, nurse coaching and peer group work approach on general health parameters in elderly individuals with diabetes mellitus. Interdisciplinary group treatment was carried out by a physiotherapist, social worker, diabetes nurse, and family physician. Clinical Pilates group treatment was carried out by a physiotherapist, and nurse coaching group treatment was carried out by a diabetes nurse. Measurements of the functional capacity of the elderly were evaluated with the Lafayette manual muscle tester and the Jamar hydraulic hand grip dynamometer. A total of 48 aged people with diabetes were randomized into 4 arms. The arms were followed up for 12 weeks.

DETAILED DESCRIPTION:
In line with the global trend, the elderly population is increasing in Turkey and the prevalence of diabetes in the elderly population continues to be high. According to the results of the Turkish Diabetes Epidemiology Study (TURDEP2), diabetic patients over the age of 65 constitute approximately 40% of all diabetics. Diabetes in an older person also increases the risk of developing frailty syndrome, which is associated with reduced muscle strength, reduced muscle quality and loss of muscle mass and accelerated aging. Muscle strength and function are reduced in diabetic patients with type 2 diabetes compared to healthy, non-glycemic individuals, with an increase in BMI and a decrease in muscle quality, when estrogen drops, especially in menopausal women. However, people with T2D may have an increased risk of falls and fractures, which may be partly explained by a decrease in muscle mass. Limited mobility can have a major impact on the individual's independence when basic daily activities like getting up from the chair, climbing stairs, and grocery shopping are disrupted for the elderly person. Decreased muscle strength can be an important factor in this loss of mobility.

In addition to physical changes, diabetes in older people also leads to emotional, mental and social difficulties and conflicts. Negative experiences such as anxiety, depression, tension and lack of social support in individuals with diabetes have bad consequences on diabetes, exacerbate the disease and increase the burden of the disease on the individual. According to the preliminary findings of the National Burden of Disease Research performed in Turkey, it has been reported that there has been a 60% increase in the burden of illness related to diabetes and that it ranks first among the burden-causing diseases. In line with all these results, a holistic approach to the phenomenon of diabetes will provide holistic interventions for the multiple effects of diabetes. However, interventions about diabetes management for the diabetic elderly are limited in the literature. Many studies have been conducted with diabetic elderly people. However, this study is the first study that includes an interdisciplinary group study for diabetic elders. The present study was organized to assess the effectiveness of these practices of an interdisciplinary care approach on the general health parameters of elderly individuals with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* individuals who were independently mobile,
* had been diagnosed with Type 2 Diabetes for a minimum of six months,
* had no serious complications or mental health issues,
* participated in regular medical check-ups,
* had no communication problems,
* agreed to participate in the study voluntarily
* aged 65 years or older.

Exclusion Criteria:

* older adults with a standardized mini-mental state examination (MMSE) score below 17
* older adults with serious complications that prevented them from participating in group activities

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Geriatric Anxiety Inventory | From enrollment to the end of treatment at 12 weeks.
  The scale's main feature is its ability to differentiate between anxious and non-anxious groups, as well as between those with and without generalised anxiety disorder. The Turkish version of the Geriatric Anxiety Inventory was used. Scores obtained from the scale range from 0 to 20. Higher scores indicate higher anxiety levels in older individuals.
Glycosylated hemoglobin | From enrollment to the end of treatment at 12 weeks.
  The glycosylated hemoglobin level is measured as a percentage according to the reference protocol of the International Federation of Clinical Chemistry. Blood samples from each patient were collected in the morning after fasting, with glycosylated hemoglobin level measurements taken one week before and again at the end of the 12-week period.
Berg Balance Scale | From enrollment to the end of treatment at 12 weeks.
  The Berg Balance Scale is a 14-item scale that quantitatively evaluates balance and fall risk. Performance is directly observed. Scores of 0 to 20 represent a lack of balance, 21 to 40 indicate acceptable balance and 41 to 56 show good balance. This scale can be used to evaluate both static and dynamic balance
Yesavage Geriatric Depression Scale | From enrollment to the end of treatment at 12 weeks.
  The scale developed by Yesavage et al., consists of 30 questions and is used as a basic screening criterion for major and minor depression. Data obtained using the Yesavage Geriatric Depression Scale were categorized as follows: 'no depression' for individuals with a score below 11; 'probable depression' for individuals with a score between 12 and 14; and 'depression' for individuals with a score of 14 or above
Type 2 Diabetes Self-Management Scale | From enrollment to the end of treatment at 12 weeks
  The scale allows for individualized assessments of lifestyle, blood glucose management and healthcare utilisation in people with type 2 Diabetes. The scale consists of 19 items across three dimensions. The healthy lifestyle behaviours subscale contains 11 items; the blood glucose management subscale contains four items; and the utilizing health services subscale contains four items
Elderly Diabetes Burden Scale | From enrollment to the end of treatment at 12 weeks.
  Araki et al. developed the scale for assessing diabetic-specific psychological aspects with 6 subscales (symptom burden, dietary restrictions, social burden, worry about diabetes, treatment dissatisfaction, and burden by tablets or insulin). The total score range for this scale is 18-88. Validity and reliability in Turkish were examined by Usta and Esen in 2012. An increase in scale scores indicates an increase in the burden in that area, and a decrease in scores indicates a low burden in that area. The Cronbach alpha coefficient for the scale was found to be 0.92
30 Seconds Sit to Stand Test | From enrollment to the end of treatment at 12 weeks.
  In the study, the 30 second sit-stand test was used, which evaluates lower body strength and endurance in older adults. Protocol developed by Rikli and Jones to determine the physical fitness levels of older adults between the ages of 60-94. The patient is asked to sit and then stand unaided for 30 seconds, and performing less than 8 repetitions is a risk indicator
Timed Up&Go Test | From enrollment to the end of treatment at 12 weeks.
  The Timed Up&Go Test includes independent measures of mobility and functional ability, including standing up from a chair, walking, turning, stopping, and sitting again. The person is asked to get up from the chair they are sitting in, walk 3 meters, come back and sit on the chair again, and the elapsed time is recorded
Gait speed measurement | From enrollment to the end of treatment at 12 weeks.
  Participants were asked to walk along a 4-metre track at their normal speed. This is an effective way of determining a person's physical function. Those who generally walk faster than 1 m/s tend to have a better functional status, a lower risk of health problems, and a higher survival rate
Hand Grip Strength | From enrollment to the end of treatment at 12 weeks.
  Muscle strength was evaluated through handgrip measurements using a handheld dynamometer (TKK 5001. Grip-A; Takei. Tokyo. Japan). Each participant completed three maximal grip trials with the left hand, followed by three with the right, with 1-min rest intervals between attempts. The test is a determinant of age-related decline in physical function
Strength of Upper/Lower Limbs | From enrollment to the end of treatment at 12 weeks.
  The handheld dynamometer (HHD), which measures isometric muscle strength, is a simple to use, easy to carry, inexpensive and light device. Quadriceps femoris, hamstring, tibialis anterior, iliopsoas, gluteus medius, biceps brachii, and shoulder abductor muscles evaluated with a handheld dynamometer

OTHER OUTCOMES:
The Standardized Mini Mental State Examination | to enrollment of participants in the enrollment session.
  The Standardized Mini Mental State Examination assesses memory, attention, orientation, language, calculation, recall, motor function, and perception. A validity and reliability study of the test was conducted in Turkey by Güngen et al. in 2002.

CONTACTS AND LOCATIONS:
Overall Officials: Huri Seval Gönderen Çakmak, Phd, Study Director — Çankırı Karatekin University
Locations (1):
- Çankırı Karatekin University Eldivan Vocational School of Health Services, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be added to the university's library and researchers can reach If they login to library's webpage. https://kutuphane.karatekin.edu.tr/.